CLINICAL TRIAL: NCT06721325
Title: EFFECTIVENESS of THERAPEUTIC EDUCATION in the PREVENTION and MANAGEMENT of SEXUAL DYSFUNCTIONS in WOMEN SURVIVORS of SEXUAL VIOLENCE and FEMALE GENITAL MUTILATION: RANDOMIZED CLINICAL TRIAL
Brief Title: THERAPEUTIC EDUCATION of SEXUAL DYSFUNCTIONS in WOMEN SURVIVORS of SEXUAL VIOLENCE and FEMALE GENITAL MUTILATION
Acronym: TESDSV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Full professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFM_SMP2024
Record Dates: First submitted 2024-07-17; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Sexual Abuse of Adult (If Focus of Attention is on Victim); Sexual Dysfunction Female; Female Genital Mutilation
Keywords: sexual violence; female genital mutilation; therapeutic education; physiotherapy
MeSH Terms: interventions — Physical Therapy Modalities; Psychotherapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL (Experimental): Psychotherapy, legal advice and physiotherapy intervention
  Interventions: Behavioral: THERAPEUTIC EDUCATION IN PHYSIOTHERAPY; Behavioral: Psychotherapy and legal advice
- CONTROL (Active Comparator): Psychotherapy and legal advice
  Interventions: Behavioral: Psychotherapy and legal advice

INTERVENTIONS:
Behavioral: THERAPEUTIC EDUCATION IN PHYSIOTHERAPY — Educational program of physiotherapy for women survivors of sexual violence and female genital mutilation.
  Arms: EXPERIMENTAL
Behavioral: Psychotherapy and legal advice — Usual psychological and legal advice therapy for this population

SUMMARY:
Violence against women is a problem that affects women all over the planet, causing physical, emotional, and other repercussions for its survivors. Pelvic floor dysfunctions, especially female sexual dysfunctions, are among the most common physical consequences for women who have suffered sexual violence or female genital mutilation. Pelvic floor physiotherapy is the first-line treatment for these dysfunctions, with therapeutic education being one of its main strategies due to its importance in the cognitive approach and for promoting patient adherence to the proposed treatments. Women who are survivors of sexual violence and female genital mutilation, being at risk for these disorders, express the need to receive information about these dysfunctions and their possible treatments. However, it has been shown that their knowledge in this regard is limited. Therefore, a project is proposed with the objective of determining the effectiveness of an intervention based on therapeutic education in the prevention and management of sexual dysfunctions secondary to sexual violence or female genital mutilation. A group educational program is proposed, which allows survivor women to address these dysfunctions in a non-invasive way. Six sessions are planned to promote the development of various competencies: communicating their needs, integrating knowledge about their health problem, identifying and analyzing, decision-making and know-how, problem-solving, using healthcare resources and asserting their rights. This will provide these women a safe space to share their experiences, learn to manage them, acquire knowledge about the pelvic floor, related dysfunctions and their treatment, as well as self-efficacy tools for dealing with sexual dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

Women who have suffered sexual assault:

* Aged 18 and older
* No severe psychiatric disorders or any other condition that prevents them from answering questions and questionnaires
* Emotionally prepared to address the affected physical and sexual sphere

Women who have undergone Female Genital Mutilation:

* Aged 18 and older
* No severe psychiatric disorders or inability to answer questions and questionnaires
* Emotionally prepared to address the affected physical and sexual sphere

Exclusion Criteria:

* Women who have suffered sexual assaults in the context of trafficking of women and girls for sexual exploitation.
* Women who have difficulty understanding the Spanish language.
* Women who are not psychologically prepared to address their sexuality.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | Before intervention (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Assessed using the Spanish version of the FSFI. The FSFI is a 19-item questionnaire that evaluates sexual function across six domains: desire, arousal, lubrication, orgasm, satis-faction, and pain. Each domain is scored from 0 to 5, with higher scores indicating better sexual function. The total FSFI score ranges from 2 to 36, with higher scores reflecting improved sexual function.

SECONDARY OUTCOMES:
Treatment Satisfaction | After completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1
  Satisfaction with the treatment will be assessed using a numerical verbal scale ranging from 0 to 10, where 0 represents no satisfaction and 10 indicates ex-cellent satisfaction. This evaluation will begin with assessment A1.

IPD SHARING:
Plan to Share IPD: No